CLINICAL TRIAL: NCT04529200
Title: Effects of Comprehensive Fall Prevention Protocol (CARE: Cognitive-Aerobic-Resistance-Exer-gaming) on Mobility Level in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, imran rafiq, Dr Imran Rafiq, Isra University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1502-PHD-004
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Fall Injury; Fall Patients; Geriatric Fall; Physical Therapy; Balance Traiing
Keywords: geriatric; fall; balance training

STUDY DESIGN:
Intervention Model Description: Total 40 patients fulfilling the inclusion criteria will be included in this study. Treatment will be given 3 times a week for 24 weeks by researcher with each session lasting for 40 to 45 Minutes. Assessment will then be done at baseline, after 04, 08, 12 and 24 weeks.
Who Masked: Participant, Care Provider
Masking Description: double blinded randomization as assessor and patient both were unaware
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. Comprehensive fall prevention protocol group (CARE) (Experimental): every week protocol change for every patient according to 1 repetition maximum
  Interventions: Other: electrotherapy treatment
- 2. Conventional balance training group (Active Comparator): conventional protocol commonly used for rehabilitation
  Interventions: Other: electrotherapy treatment

INTERVENTIONS:
Other: electrotherapy treatment — physical therapy management like EMS IFT

SUMMARY:
Lack of research oriented health care facilities especially rehabilitation department in Pakistan. 30-50 % of population of age 65 years and above have some problems with balance (3) and 75 % of people aging 70 years and above have poor balance which leads to fall related injuries (5). So fall and related injuries are major problem in this age group. All studies conducted so far addresses only one or two aspects of balance training not to all. This study will address all the aspects and develop a comprehensive balance training protocol and will try to contribute to this under research area.

DETAILED DESCRIPTION:
Lack of research oriented health care facilities especially rehabilitation department in Pakistan. 30-50 % of population of age 65 years and above have some problems with balance (3) and 75 % of people aging 70 years and above have poor balance which leads to fall related injuries (5). So fall and related injuries are major problem in this age group. All studies conducted so far addresses only one or two aspects of balance training not to all. This study will address all the aspects and develop a comprehensive balance training protocol and will try to contribute to this under research area.

Cost effective treatment for patients. To meet the expectation of patient to improve their quality of life and improvement of their satisfactory level. It will be interesting for patient to visualize the activity patient is performing and comparison of effectiveness of comprehensive fall prevention protocol with traditional balance training.

It will reduce the occurrence of fall episodes and hence reduce the cost to treat these fall and fall related injuries. Older adult will be less dependent, and more mobile and contributing member of the community.

Objectives

The objectives of the study are:

1. To compare the effect of comprehensive fall prevention protocol (CARE) on fall risk as compared to conventional training in elderly.
2. To compare the effect of comprehensive fall prevention protocol (CARE) on Mobility Level as compared to conventional training in elderly.
3. To compare the effect of comprehensive fall prevention protocol (CARE) on Wii Fit balance as compared to conventional training in elderly.
4. To compare the effect of comprehensive fall prevention protocol (CARE) on Dynamic Balance as compared to conventional training in elderly.
5. To compare the effect of comprehensive fall prevention protocol (CARE) on Quality of life as compared to conventional training in elderly.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of age 60 -80 years
* Either gender
* Berg balance score between 20-40

Exclusion Criteria:

* • Musculoskeletal conditions (fractures, severe arthritis)

  * Neurological conditions like Epilepsy, Parkinson,
  * Alzheimer's, Impaired cognition
  * Other systemic diseases or co-morbidities

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-05 (Actual); Primary Completion 2020-11-10 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Elderly mobility scale | 8 week
  questionaire used to evaluate condition of elders
Timed Up and go test (TUG) | 8 week
  questionaire used to evaluate mobility
Berg Balance Test | 8 week
  questionaire used to evaluate balance
Activities of Balance Confidence | 8 week
  questionaire used to evaluate balance
Fullerton Advanced Balance (FAB) Scale | 8 week
  questionaire used to evaluate function of balance in older adult
Functional reach test | 8 week
  This test measures the distance between the length of an outstretched arm in a maximal forward reach from a standing position,while maintaining a fixed base of support.
Dynamic gait index | 8 week
  The Dynamic Gait Index (DGI) was developed as a clinical tool to assess gait, balance and fall risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Isra University, Islamabad, Capital, Pakistan